CLINICAL TRIAL: NCT03810300
Title: Sustainability of Impacts of Cash Transfers, Food Transfers, and Behavior Change Communication in Bangladesh: Transfer Modality Research Initiative
Brief Title: Sustainability of Impacts of Cash Transfers, Food Transfers, and Behavior Change Communication in Bangladesh
Acronym: TMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: Cornell University (Other); Data Analysis and Technical Assistance Ltd (Unknown); World Food Programme, Bangladesh (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 12835
Record Dates: First submitted 2018-05-14; First posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Food Security; Poverty; Child Nutrition; Child Development; Intimate Partner Violence; Gender Dynamics
Keywords: Cash transfers; Food transfers; Behavior change communication; Sustainability; Social protection; Nutrition; Gender
MeSH Terms: conditions — Coitus | interventions — Food

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cash transfer (Experimental): 1500 taka ($18.75) per household distributed monthly
  Interventions: Other: Cash transfer
- Food transfer (Experimental): 30 kg rice, 2 kg lentils, and 2 kg micro-nutrient fortified cooking oil per household distributed monthly
  Interventions: Other: Food transfer
- Food and cash transfer (Experimental): 15 kg of rice; 1 kg of lentils and 1 kg of micronutrient fortified cooking oil and 750 taka cash per household, distributed monthly
  Interventions: Other: Food and cash transfer
- Cash transfer + nutrition BCC (Experimental): 1500 taka ($18.75) per household distributed monthly. Nutrition behavior change communication (weekly, one-hour group-based meetings on maternal and child nutrition, sanitation and health knowledge, attitudes and practice; twice-a-month home visits; monthly community meetings).
  Interventions: Other: Cash transfer; Behavioral: Nutrition behavior Communication Change (BCC)
- Food transfer + nutrition BCC (Experimental): 30 kg rice, 2 kg lentils, and 2 kg micro-nutrient fortified cooking oil per household distributed monthly. Nutrition behavior change communication (weekly, one-hour group-based meetings on maternal and child nutrition, sanitation and health knowledge, attitudes and practice; twice-a-month home visits; monthly community meetings).
  Interventions: Other: Food transfer; Behavioral: Nutrition behavior Communication Change (BCC)
- Control (Experimental): No transfer, no behavior change communication
  Interventions: Other: Control

INTERVENTIONS:
Other: Cash transfer — 1500 taka ($18.75) per household distributed monthly
  Arms: Cash transfer; Cash transfer + nutrition BCC
Other: Food transfer — 30 kg rice, 2 kg lentils, and 2 kg micro-nutrient fortified cooking oil per household distributed monthly
  Arms: Food transfer; Food transfer + nutrition BCC
Other: Food and cash transfer — 15 kg of rice, 1 kg of lentils, and 1 kg of micronutrient-fortified cooking oil, and 750 taka cash per household, distributed monthly
  Arms: Food and cash transfer
Behavioral: Nutrition behavior Communication Change (BCC) — Weekly, group-based, one-hour meetings on maternal and child nutrition, sanitation and health knowledge, attitudes and practice; twice-a-month home visits; monthly community meetings
  Arms: Cash transfer + nutrition BCC; Food transfer + nutrition BCC
Other: Control — No transfer, no behavior change communication
  Arms: Control

SUMMARY:
This study assesses the sustainability of impacts, 4 years post-program, from a pilot safety net program that was implemented from May 2012-April 2014. The intervention, called the Transfer Modality Research Initiative (TMRI), was assigned following a cluster-randomized controlled trial design in two zones of Bangladesh (north and south). Intervention arms were assigned at the village level, where arms were as follows: (1) cash transfers [north and south]; (2) cash transfers + nutrition behavior communication change (BCC) [north only]; (3) food transfers [north and south]; (4) food transfers + nutrition BCC [south only]; (4) food-cash split [north and south]; and (5) control [north and south]. Within treatment villages, women living in very poor households were targeted to receive benefits for two years.

DETAILED DESCRIPTION:
The objective of the study is to assess, 4 years after a pilot safety net intervention ended in April 2014, the sustainability of the intervention's impacts on households, children, and women. The intervention, called the Transfer Modality Research Initiative (TMRI), was assigned following a cluster-randomized controlled trial design in two zones of Bangladesh (north and south). WFP-Bangladesh implemented the intervention, and the International Food Policy Research Institute (IFPRI) conducted the impact evaluation research. Intervention arms were assigned at the village level, where arms were as follows: (1) cash transfers [north and south]; (2) cash transfers + nutrition behavior communication change (BCC) [north only]; (3) food transfers [north and south]; (4) food transfers + nutrition BCC [south only]; (5) food-cash split [north and south]; and (5) control [north and south]. Within treatment villages, women living in very poor households were targeted to receive benefits for two years, from May 2012-April 2014. For the original impact evaluation, longitudinal data on 5000 households were collected from 2012-2015 (ClinicalTrials.gov Identifier: NCT02237144).

For the sustainability study in 2018, given available funding, the sampling frame will include 4000 households. This will include all households that were originally in the following arms: (1) cash transfers [north and south]; (2) cash transfers + nutrition BCC [north only]; (3) food transfers [north and south]; (4) food transfers + nutrition BCC [south only]; (5) control [north and south].

ELIGIBILITY:
Inclusion Criteria:

* Former participant of Transfer Modality Research Initiative study (in cash, food, cash+BCC, food+BCC, or control arms)

Exclusion Criteria:

-

Ages: 15 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 5000 (Actual)
Dates: Start 2012-04-15 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Food Consumption Score | After 4 years post-intervention
  The Food Consumption Score, as defined by the World Food Programme, is calculated as the number of food groups consumed by the household in the previous 7 days, weighted by each food group's nutritional value and frequency of consumption. Scale range is 0 to 112, with higher values reflecting higher food consumption.
Child height-for-age z-score | After 4 years post-intervention
  Calculated using the 2006 WHO growth reference. This is a continuous measure that represents the number of standard deviations from the mean among comparable children in the WHO growth reference.
Prevalence of physical intimate partner violence | After 4 years post-intervention
  Prevalence of any physical intimate partner violence in the past 12 months measured using the WHO Violence Against Women instrument

SECONDARY OUTCOMES:
Household dietary diversity | After 4 years post-intervention
  Measured by counting the number of food groups consumed by the household
Value of total household consumption | After 4 years post-intervention
  Aggregate value of household food and non-food consumption expenditures. This is a continuous measure calculated from household survey responses on consumption behavior, using the methodology and questionnaire modules described in Deaton and Zaidi (2002). Citation: A.Deaton,, and S. Zaidi. 2002. "Guidelines for Constructing Consumption Aggregates for Welfare Analysis." Washington, DC : World Bank.
Value of household food consumption | After 4 years post-intervention
  Value of household food consumption expenditures. This is a continuous measure calculated from household survey responses on consumption behavior, using the methodology and questionnaire modules described in Deaton and Zaidi (2002). Citation: A.Deaton,, and S. Zaidi. 2002. "Guidelines for Constructing Consumption Aggregates for Welfare Analysis." Washington, DC : World Bank.
Value of household non-food consumption | After 4 years post-intervention
  Value of household non-food consumption expenditures. This is a continuous measure calculated from household survey responses on consumption behavior, using the methodology and questionnaire modules described in Deaton and Zaidi (2002). Citation: A.Deaton,, and S. Zaidi. 2002. "Guidelines for Constructing Consumption Aggregates for Welfare Analysis." Washington, DC : World Bank.
Household food insecurity | After 4 years post-intervention
  Measured using the Household Food Insecurity Access Scale. Scale range is 0 to 27, with higher values reflecting higher food insecurity.
Value of household labor income | After 4 years post-intervention
  Value of annual labor income over all household members
Value of household non-labor income | After 4 years post-intervention
  Value of annual non-labor income over all household members
Value of household asset ownership | After 4 years post-intervention
  Total value of all assets owned
Household land ownership | After 4 years post-intervention
  Area of land owned
Housing quality: interviews | After 4 years post-intervention
  Quality of housing stock. This is measured using a module developed for the study context, and information is collected through household enumerator observation during interviews.
Maternal nutrition knowledge score | After 4 years post-intervention
  Number answered correctly on a test of maternal knowledge regarding infant and young child feeding practices developed for the survey, based on the curriculum of training sessions in the intervention.
Maternal infant and young child feeding practices | After 4 years post-intervention
  Maternal adherence to WHO-recommended infant and young child feeding practices
Child score on Raven's Progressive Matrices | After 4 years post-intervention
  Measured using Raven's Progressive Matrices set A and set B. This is constructed following the test's protocol for scoring.
Child score on Early Grade Reading Assessment | After 4 years post-intervention
  Measured using Early Grade Reading Assessment adapted to local context. This is constructed following the test's protocol for scoring.
Child score on Early Grade Mathematics Assessment | After 4 years post-intervention
  Measured using Early Grade Mathematics Assessment adapted to local context. This is constructed following the test's protocol for scoring.
Child score on Strengths and Difficulties Questionnaire | After 4 years post-intervention
  Measured using Strengths and Difficulties Questionnaire, part of the Development and Well-Being Assessment family of mental heath measures. This is constructed following the test's protocol for scoring.
Child weight-for-height z-score | After 4 years post-intervention
  Calculated using the 2006 WHO growth reference. This is a continuous measure that represents the number of standard deviations from the mean among comparable children in the WHO growth reference.
Prevalence of child stunting | After 4 years post-intervention
  Calculated using the 2006 WHO growth reference
Prevalence of child wasting | After 4 years post-intervention
  Calculated using the 2006 WHO growth reference
Child illness | After 4 years post-intervention
  Mother's report of child illness in previous 2 weeks
Parental interaction with child | After 4 years post-intervention
  Time spent on child stimulation activities in previous 7 days, measured using modules developed for the survey
Parental discipline of the child | After 4 years post-intervention
  Disciplinary measures used in the past month, measured using modules developed for the survey
Community norms on gender | After 4 years post-intervention
  Community leaders' attitudes toward gender, measured using modules developed for the survey
Prevalence of emotional violence | After 4 years post-intervention
  Prevalence of any emotional intimate partner violence in the past 12 months measured using the WHO Violence Against Women instrument
Prevalence of controlling behaviors | After 4 years post-intervention
  Prevalence of any controlling behaviors in the past 12 months measured using the WHO Violence Against Women instrument
Prevalence of individual acts of intimate partner violence | After 4 years post-intervention
  Prevalence of individual acts of intimate partner violence in the past 12 months measured using the WHO Violence Against Women instrument
Individual decisionmaking | After 4 years post-intervention
  Measured using men's and women's decisionmaking modules adapted from pro-WEAI
Individual asset ownership | After 4 years post-intervention
  Measured using men's and women's asset ownership modules developed for the survey
Individual mobility | After 4 years post-intervention
  Measured using men's and women's mobility modules adapted from pro-WEAI
Individual labor force participation | After 4 years post-intervention
  Measured using men's and women's labor modules developed for the survey
Individual attitudes toward gender and intimate partner violence | After 4 years post-intervention
  Measured using men's and women's attitudes toward gender and intimate partner violence modules developed for the survey
Individual social capital | After 4 years post-intervention
  Measured using men's and women's social capital modules developed for the survey
Individual stress | After 4 years post-intervention
  Measured using men's and women's Perceived Stress Scale scores
Individual depression | After 4 years post-intervention
  Measured using men's and women's Patient Health Questionnaire-9 Depression Test scores
Individual aspirations | After 4 years post-intervention
  Measured using men's and women's aspirations modules developed for the survey
Spousal relationship | After 4 years post-intervention
  Measured using men's and women's relationship modules developed for the survey

CONTACTS AND LOCATIONS:
Overall Officials: Akhter Ahmed, PhD, Principal Investigator — International Food Policy Research Institute; Shalini Roy, PhD, Principal Investigator — International Food Policy Research Institute; John Hoddinott, DPhil, Principal Investigator — Cornell University; Melissa Hidrobo, PhD, Principal Investigator — International Food Policy Research Institute